CLINICAL TRIAL: NCT02385253
Title: Training Primary Care Physicians to Perform Melanoma Opportunistic Surveillance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, June Robinson, Professor of Dermatology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: STU00082564
Record Dates: First submitted 2015-02-25; First posted 2015-03-11 (Estimated); Last update posted 2018-06-07 (Actual); Status verified 2017-09

CONDITIONS: Melanoma; Nevi; Skin Moles
Keywords: Training; Primary Health Care; Skin Cancer; Primary Care Physicians; Surveillance; Education
MeSH Terms: conditions — Melanoma; Nevus; Skin Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Educational training program (Active Comparator): PCPs randomized to the intervention group will receive the educational training program at the beginning of the study, extending over a maximum of five months.
  Interventions: Behavioral: Educational training program
- Control (No Intervention): PCPs randomized to the control group will have the option of receiving the educational training program at the end of the study.

INTERVENTIONS:
Behavioral: Educational training program — The educational training program (intervention) consists of four sequential phases:
  1. Knowledge Acquisition
  2. Skills Assessment
  3. Deliberate Practice
  4. Clinical Proficiency
  Arms: Educational training program

SUMMARY:
This is a four-phase educational intervention for primary care practitioners (PCPs) to perform opportunistic melanoma surveillance. Based on prior research, the investigator will develop an interactive melanoma early detection skills training program for PCPs according to the principals of mastery learning. The proposed educational intervention will improve practicing PCPs' knowledge, competence, confidence, and diagnostic performance regarding pigmented lesions and attitude concerning importance of skin surveillance. In addition, this research aims to examine the clinical proficiency of PCPs regarding pigmented lesions. The proposed educational intervention will reduce the percentage of benign lesions referred to dermatology.

DETAILED DESCRIPTION:
Cutaneous melanoma is considered a potentially curable disease if detected early. Primary care physicians (PCPs) are well positioned to detect early melanomas by performing opportunistic melanoma surveillance on the at-risk population during physical examination. Opportunistic surveillance means physician performance of visual inspection of skin exposed during your physical examination focused on the presenting condition. Opportunistic surveillance requires skills in both visual inspection of the skin and with magnification of the skin by a hand-held device, a dermoscope. (This research aims to 1) develop an easily disseminated, interactive melanoma early detection skills training program for PCPs and to 2) to examine the clinical proficiency of PCPs regarding pigmented lesions.

The knowledge to be gained by PCPs is essential to the development and successful introduction of a method for physicians to learn how to perform opportunistic surveillance for melanoma. By evaluating means of encouraging and facilitating opportunistic surveillance for melanoma, an educational program may eventually be brought into widespread use in training PCPs.

In addition to a Pre-training Test and Post-training Test, each of the phases of the educational training program is described below:

1. Knowledge Acquisition The Knowledge Acquisition phase will be delivered via personal computer/tablet. It will take about one hour to complete. The one-hour course consists of case histories and videos in which the following are presented: 1) threshold rules of visual inspection, 2) benefit of magnification with dermoscopy to assist with diagnosis, and 3) demonstration of the 3-point checklist of dermoscopy.
2. Skills Assessment The Skills Assessment phase will be delivered via smartphone. The program may be intermittently accessed taking up to two weeks to complete. The PCP will be asked to review and make simulated management decisions on 20 case vignettes with clinical images of body surfaces and dermoscopy of individual lesions. Clinical practice will be simulated with the requirement that you make a decision to refer to dermatology or a decision that a referral is not needed. If a biopsy is performed in the case vignette, the pathology report will be provided, and the PCP will be asked the next step in the patient's care. Performance feedback will be provided.
3. Deliberate Practice The Deliberate Practice phase will be delivered via smartphone. It will take between 1-8 weeks to complete. The PCP will be asked to review additional cases with visual inspection and dermoscopy to improve aspects of your performance that have demonstrated weakness. Individual strengths and weaknesses will be assessed, and personalized feedback will be provided. After achieving competency with the simulated cases, the research staff will provide the PCP with a DermScope device (a smartphone fitted with a dermoscope) to use in the next phase.
4. Clinical Proficiency The Clinical Proficiency phase will take place in the clinical practice of the PCP over the course of 1-8 weeks. The PCP will be asked to use the DermScope to capture and transmit at least 12 lesions. Informed consent will be obtained from each patient prior to obtaining the non-identifying images. During image capture, each photograph is marked by the DermScope program with the date, time, and the clinical assessment form (CAF). The image will be transmitted to the teleconsultant (PI), who will assign a unique identification number to the image and the data. The PI will render an opinion within 72 hours regarding the need to refer the patient to dermatology or reassure the patient. The PCP will be asked to make a decision regarding the management of the patient and communicate this decision as needed to the patient.

ELIGIBILITY:
Inclusion Criteria for PCPs:

* is a practicing PCP in the section of General Internal Medicine of Northwestern Medicine

Exclusion Criteria for PCPs:

* is NOT a practicing PCP in the section of General Internal Medicine of Northwestern Medicine

Inclusion Criteria for Patients providing lesions to be photographed:

* is a patient of a PCP enrolled in the study
* is at least 18 years old
* able to read at a 6th grade level or higher

Exclusion Criteria for Patients providing lesions to be photographed:

* is NOT a patient of a PCP enrolled in the study
* under 18 years of age
* unable to read at a 6th grade level

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2015-09-15 (Actual); Primary Completion 2017-07-23 (Actual); Study Completion 2017-07-23 (Actual)

PRIMARY OUTCOMES:
Change from baseline performance at 5 months (difference-in-difference) | Baseline and 5 months
  The difference-in-difference (DID) approach will be used to test the hypothesis that the educational intervention improved knowledge, attitude concerning importance of skin exam, competence, confidence, and diagnostic performance. The difference-in-difference estimator compares outcomes between pre-tests and post-tests between PCPs who received the educational intervention and those who did not.
  Each PCP will be the unit of observation. We will choose an appropriate functional form for each outcome.For each outcome, a DID estimator that is significant at p < 0.05 will support the hypothesis that the educational intervention improved outcomes. This analysis will be repeated for each of the five outcomes. We will use the Bonferroni correction for multiple comparisons.

SECONDARY OUTCOMES:
Change in number of pigmented lesions referrals from three months prior and three months post randomization (Difference-in-Difference estimator) | Three months prior randomization, Three months post intervention
  The difference-in-difference (DID) approach will be used to test the hypothesis that the intervention reduced referrals of benign lesions. The model will be estimated using a random effects logistic regression to account for clustering due to repeated measures for each PCP (about 8 referrals before randomization and another 8 after the intervention). A 95% confidence interval for the odds ratio of α3 that falls below one will support the hypothesis.

CONTACTS AND LOCATIONS:
Overall Officials: June K Robinson, MD, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Northwestern Medicine: Division of General Internal Medicine and Geriatrics, Chicago, Illinois
  - Northwestern University Feinberg School of Medicine Department of Dermatology, Chicago, Illinois

REFERENCES:
- [Background] Robinson JK, Jain N, Marghoob AA, McGaghie W, MacLean M, Gerami P, Hultgren B, Turrisi R, Mallett K, Martin GJ. A Randomized Trial on the Efficacy of Mastery Learning for Primary Care Provider Melanoma Opportunistic Screening Skills and Practice. J Gen Intern Med. 2018 Jun;33(6):855-862. doi: 10.1007/s11606-018-4311-3. Epub 2018 Feb 5. PMID 29404948
- [Background] Robinson JK, MacLean M, Reavy R, Turrisi R, Mallett K, Martin GJ. Dermoscopy of Concerning Pigmented Lesions and Primary Care Providers' Referrals at Intervals After Randomized Trial of Mastery Learning. J Gen Intern Med. 2018 Jun;33(6):799-800. doi: 10.1007/s11606-018-4419-5. No abstract available. PMID 29637481